CLINICAL TRIAL: NCT00298623
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of XP13512 in Patients With Restless Legs Syndrome.
Brief Title: XP13512 (GSK1838262) Versus Placebo in Patients With Restless Legs Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Cheri Hudson; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110963
Record Dates: First submitted 2006-02-28; First posted 2006-03-02 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2011-05

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: placebo
- XP13512 (GSK1838262) (Experimental)
  Interventions: Drug: XP13512 (GSK1838262)

INTERVENTIONS:
Drug: XP13512 (GSK1838262)
  Arms: XP13512 (GSK1838262)
Other: placebo
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to assess the efficacy of XP13512 taken once daily compared to placebo for the treatment of patients suffering from Restless Legs Syndrome (RLS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary RLS, based on the International RLS Study Group Diagnostic Criteria.
* History of RLS symptoms at least 15 nights in the prior month or, if on treatment, this frequency of symptoms before treatment was started;
* Documented RLS symptoms for at least 4 of the 7 consecutive evenings/nights during the Baseline study period;
* Total RLS severity score of 15 or greater on the International Restless Legs Syndrome Study Group Rating Scale (IRLS rating scale) at Visit 1 and at Visit 2;
* Discontinuation of dopamine agonists and/or gabapentin at least 2 weeks prior to Baseline;
* Discontinuation of other treatments for RLS (e.g., opioids, benzodiazepines) at least 2 weeks prior to Baseline;
* If female of child-bearing potential, the subject must agree to use clinically accepted birth control through completion of the study;
* Body Mass Index of 34 or below;
* Estimated creatinine clearance of at least 60 mL/min;

Exclusion Criteria:

* A sleep disorder (e.g., sleep apnea) that may significantly affect the assessment of RLS;
* Neurologic disease or movement disorder (e.g., diabetic neuropathy, Parkinson's Disease, Multiple Sclerosis, dyskinesias, and dystonias);
* Abnormal laboratory results, electrocardiogram (ECG) or physical findings;
* Pregnant or lactating women;
* Women of childbearing potential who are not practicing an acceptable method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2006-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The change from baseline to the end of treatment in International Restless Legs Syndrome (IRLS) rating scale score. | 12-week treatment period
The proportion of subjects at the end of treatment who are "much improved" or "very much improved" on the Investigator-rated CGI of Improvement | 12-week treatment period

SECONDARY OUTCOMES:
Onset of efficacy. Subjective measures of sleep. | 12-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Kushida CA, Walters AS, Becker P, Thein SG, Perkins AT, Roth T, Canafax D, Barrett RW; XP021 Study Group. A randomized, double-blind, placebo-controlled, crossover study of XP13512/GSK1838262 in the treatment of patients with primary restless legs syndrome. Sleep. 2009 Feb;32(2):159-68. doi: 10.1093/sleep/32.2.159. PMID 19238802
- [Derived] Ahmed M, Hays R, Steven Poceta J, Jaros MJ, Kim R, Shang G. Effect of Gabapentin Enacarbil on Individual Items of the International Restless Legs Study Group Rating Scale and Post-sleep Questionnaire in Adults with Moderate-to-Severe Primary Restless Legs Syndrome: Pooled Analysis of 3 Randomized Trials. Clin Ther. 2016 Jul;38(7):1726-1737.e1. doi: 10.1016/j.clinthera.2016.05.008. Epub 2016 Jun 7. PMID 27288210
- [Derived] Avidan AY, Lee D, Park M, Jaros MJ, Shang G, Kim R. The Effect of Gabapentin Enacarbil on Quality of Life and Mood Outcomes in a Pooled Population of Adult Patients with Moderate-to-Severe Primary Restless Legs Syndrome. CNS Drugs. 2016 Apr;30(4):305-16. doi: 10.1007/s40263-016-0329-4. PMID 27067343
- [Derived] Ondo WG, Hermanowicz N, Borreguero DG, Jaros MJ, Kim R, Shang G. Effect of prior exposure to dopamine agonists on treatment with gabapentin enacarbil in adults with moderate-to-severe primary restless legs syndrome: pooled analyses from 3 randomized trials. J Clin Mov Disord. 2015 Mar 30;2:9. doi: 10.1186/s40734-015-0018-3. eCollection 2015. PMID 26788345
- [Derived] Canafax DM, Bhanegaonkar A, Bharmal M, Calloway M. Validation of the post sleep questionnaire for assessing subjects with restless legs syndrome: results from two double-blind, multicenter, placebo-controlled clinical trials. BMC Neurol. 2011 Apr 28;11:48. doi: 10.1186/1471-2377-11-48. PMID 21527006